CLINICAL TRIAL: NCT01480232
Title: Proof-of-Concept Study of EVP-6124, an Alpha-7 Nicotinic Acetylcholine Receptor Agonist, Versus Placebo in Subjects With Nicotine Dependence
Brief Title: A Safety and Cognitive Function Study of EVP-6124 Versus Placebo in Subjects With Nicotine Dependence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been put on clinical hold by FDA
Sponsor: A. Eden Evins (Other)
Collaborators: FORUM Pharmaceuticals Inc (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, A. Eden Evins, Director, Center for Addiction Medicine Massachusetts General Hospital, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EVP-6124-014; 1R01DA030992-01 (NIH)
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-02

CONDITIONS: Nicotine Dependence; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — 7-chloro-N-quinuclidin-3-yl-benzo(b)thiophene-2-carboxamide; Exercise; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EVP-6124 + NicoDerm (Active) (Experimental): One EVP-6124 capsule ingested orally daily for 12 weeks (84 days) and one NicoDerm patch (Active) daily for first 6 weeks (42 days)
  Interventions: Drug: EVP-6124; Drug: NicoDerm Patch (Active); Behavioral: Brief Supportive and Behavioral Treatment
- Placebo + NicoDerm (Active) (Active Comparator): One placebo capsule ingested orally daily for 12 weeks (84 days) and one NicoDerm patch (Active) daily for first 6 weeks (42 days)
  Interventions: Drug: Placebo Capsule; Drug: NicoDerm Patch (Active); Behavioral: Brief Supportive and Behavioral Treatment
- EVP-6124 + NRT Patch (Placebo) (Experimental): One EVP-6124 capsule ingested orally daily for 12 weeks (84 days) and one NRT patch (Placebo) daily for first 6 weeks (42 days)
  Interventions: Drug: EVP-6124; Drug: NRT Patch (Placebo); Behavioral: Brief Supportive and Behavioral Treatment
- Placebo + NRT Patch (Placebo) (Placebo Comparator): One placebo capsule ingested orally daily for 12 weeks (84 days) and one NRT patch (Placebo) daily for first 6 weeks (42 days)
  Interventions: Drug: Placebo Capsule; Drug: NRT Patch (Placebo); Behavioral: Brief Supportive and Behavioral Treatment

INTERVENTIONS:
Drug: EVP-6124 — One EVP-6124 capsule ingested orally daily for 12 weeks (84 days)
  Arms: EVP-6124 + NRT Patch (Placebo); EVP-6124 + NicoDerm (Active)
Drug: Placebo Capsule — One placebo capsule ingested orally daily for 12 weeks (84 days)
  Arms: Placebo + NRT Patch (Placebo); Placebo + NicoDerm (Active)
Drug: NicoDerm Patch (Active) — One NicoDerm patch once daily for first 6 weeks (42 days). Dosage will taper from 21 mg (Weeks 1-3) to 14 mg (Weeks 4-5) to 7 mg (Week 6).
  Arms: EVP-6124 + NicoDerm (Active); Placebo + NicoDerm (Active)
Drug: NRT Patch (Placebo) — One NRT patch (Placebo) daily for first 6 weeks (42 days).
  Arms: EVP-6124 + NRT Patch (Placebo); Placebo + NRT Patch (Placebo)
Behavioral: Brief Supportive and Behavioral Treatment — Brief, standard, manualized individual cognitive behavioral therapy intervention will be based on the Freedom from Smoking curriculum from the American Lung Association.

SUMMARY:
This study is designed to evaluate the initial evidence for efficacy of the investigational medicine, EVP-6124, to improve smoking cessation outcomes with and without a standard taper of nicotine replacement therapy (NRT) in healthy nicotine dependent smokers

ELIGIBILITY:
Inclusion Criteria:

* Self-report of smoking an average of ≥10 cigarettes/day for 6 months and expired carbon monoxide (CO) ≥10 parts per million (ppm) or urine cotinine ≥ 100 ng/mL at screening or self-report of smoking an average of 5-9 cigarettes/day for 6 months and a urine cotinine ≥30ng/ml at screening
* Have a negative urine drug screen at screening
* Fertile, sexually active subjects (males and females) must use an effective method of contraception from the first dose of study drug and for 3 months after the last dose of study drug
* If female and capable of conception, must have a negative urine Human chorionic gonadotrophin (hCG) pregnancy test at screening and Day 1

Exclusion Criteria:

* Have unstable medical illness with hospitalization for treatment likely within 6 months
* Have life-threatening arrhythmia, cerebrovascular or cardiovascular event within 6 months of enrollment
* Have liver function tests elevated >2.5 times the upper limit of normal range
* Have a tumor or a seizure disorder
* Currently using other tobacco- or nicotine-containing products and unwilling to try to quit
* Have a 6-month history of substance use disorder other than nicotine or caffeine or major depressive disorder
* Have a history of multiple adverse drug reactions
* Non-response (past 3 months) to nicotine replacement therapy (NRT) >20 mg/day, bupropion >150 mg/day, or varenicline 2 mg/day for ≥4 weeks
* Use of excluded concomitant medications
* Hospitalization for any reason within 30 days of screening
* Use of any investigational drug or device within 30 days of screening
* Have clinically significant abnormal serum electrolytes
* Have insufficiently controlled diabetes mellitus
* Have renal insufficiency (serum creatinine >1.8 mg/dL)
* Malignant tumor within the last 5 years, with the exception of squamous and basal cell carcinoma or cervical carcinoma in situ
* Have a clinically significant cardiovascular abnormality on the screening EKG
* Lifetime history of schizophrenia, bipolar disorder, post-traumatic stress disorder, bulimia, organic mental disorder, dementia, pervasive developmental disorder
* Have untreated, clinically significant hypothyroidism or hyperthyroidism
* Have a positive self-report of human immunodeficiency virus infection
* Females who are pregnant or nursing
* Any experimental drug currently or within 30 days before baseline
* Have a serious risk of suicide
* Have a screening electrocardiogram (ECG) with a corrected QT (QTc) interval using Bazett's formula >450 msec for males and >470 msec for females or the presence of any clinically significant cardiac abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2011-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital; Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited using advertisements in the local media market.Those who made contact in response to advertisements spoke initially with a research coordinator who provided further information about the study, answered initial questions from the potential subject, and administered a 10-minute questionnaire assessing eligibility.
Pre-assignment Details: Prior to initiation of any study procedures, the informed consent process was conducted by a study physician who explained the study in detail making sure that the subject understood the potential risks/benefits as outlined in the consent form; 350 signed consent, 60 were found ineligible and 130 either withdrew consent or was discontinued
Groups:
- EVP-6124 + NRT Patch (Placebo): One EVP-6124 capsule ingested orally daily for 12 weeks (84 days) and one NRT patch (Placebo) daily for first 6 weeks (42 days)
  EVP-6124: One EVP-6124 capsule ingested orally daily for 12 weeks (84 days)
  NRT (nicotine replacement therapy) Patch (Placebo): One NRT patch (Placebo) daily for first 6 weeks (42 days).
  Brief Supportive and Behavioral Treatment: Brief, standard, manualized individual cognitive behavioral therapy intervention will be based on the Freedom from Smoking curriculum from the American Lung Association.
Period: Overall Study
Arm/Group | EVP-6124 + NicoDerm (Active) | EVP-6124 + NRT Patch (Placebo) | Placebo + NicoDerm (Active) | Placebo + NRT Patch (Placebo)
Started | 40 | 41 | 38 | 41
Completed | 22 | 19 | 21 | 22
Not Completed | 18 | 22 | 17 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EVP-6124 + NicoDerm (Active) | EVP-6124 + NRT Patch (Placebo) | Placebo + NicoDerm (Active) | Placebo + NRT Patch (Placebo) | Total
Number analyzed (Participants) | 40 | 41 | 38 | 41 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.63 (12.17) | 44.70 (13.06) | 44.03 (12.81) | 45.15 (11.42) | 44.30 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 13 | 17 | 58
  Male | 26 | 27 | 25 | 24 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 3 | 1 | 16
  Not Hispanic or Latino | 32 | 37 | 35 | 40 | 144
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30 | 36 | 29 | 30 | 125
  African American | 8 | 3 | 7 | 10 | 28
  Other | 2 | 2 | 2 | 1 | 7
Years of Regular Smoking [Mean (Standard Deviation); unit: years] | 23.31 (11.01) | 26.38 (13.24) | 24.89 (12.84) | 26.46 (12.17) | 25.26 (12.32)
Cigarettes Smoked Per Day [Mean (Standard Deviation); unit: cigarettes per day] | 18.53 (9.35) | 19.41 (15.09) | 22.87 (30.63) | 20.04 (13.85) | 20.21 (17.23)
Expired CO, ppm [Mean (Standard Deviation); unit: parts per million] — Measurements of CO in expired breath was the primary means of biochemical verification of smoking self-report during the study at each study visit. End-expiratory CO levels ≥10 ppm indicate current cigarette use, whereas levels of <10 ppm indicate abstinence.
  parts per million | 5.18 (4.17) | 4.29 (2.76) | 4.78 (3.46) | 4.85 (4.38) | 4.78 (3.69)
FTND Score [Mean (Standard Deviation); unit: units on a scale] — Fagerström Test for Nicotine Dependence (FTND) will determine the level of nicotine dependence. The scale score ranges from 0 to 10. An FTND score ≥6 indicates high nicotine dependence and a score of <6 indicates a low to moderate level of dependence
  units on a scale | 5.40 (2.07) | 5.34 (2.17) | 5.39 (1.94) | 5.32 (2.07) | 5.36 (2.06)

OUTCOME MEASURES:

1. Primary Outcome: Effects of EVP-6124 on 7-day Point-prevalence Smoking Abstinence
Description: Smoking abstinence is defined as a self-report of smoking no cigarettes for the past 7 days by time-line follow-back, confirmed by expired carbon monoxide (CO) <10 ppm and/or urine cotinine <50 ng/mL.
Time Frame: Week 1, 2, 4, 6, 8, 10, 12
Population: The primary smoking cessation variable is biochemically verified self-report of 7-day point prevalence abstinence at 12 weeks (end of treatment).
Measure: Number; unit: % participants with 7-Day Point Prevalen
Groups:
- EVP-6124 + NicoDerm CQ (Active): One EVP-6124 capsule ingested orally daily for 12 weeks (84 days) and one NicoDerm CQ patch (Active) daily for first 6 weeks (42 days)
  EVP-6124: One EVP-6124 capsule ingested orally daily for 12 weeks (84 days)
  NicoDerm CQ Patch (Active): One NicoDerm CQ patch once daily for first 6 weeks (42 days). Dosage will taper from 21 mg (Weeks 1-3) to 14 mg (Weeks 4-5) to 7 mg (Week 6).
  Brief Supportive and Behavioral Treatment: Brief, standard, manualized individual cognitive behavioral therapy intervention will be based on the Freedom from Smoking curriculum from the American Lung Association.
- Placebo + NicoDerm CQ (Active): One placebo capsule ingested orally daily for 12 weeks (84 days) and one NicoDerm CQ patch (Active) daily for first 6 weeks (42 days)
  Placebo Capsule: One placebo capsule ingested orally daily for 12 weeks (84 days)
  NicoDerm CQ Patch (Active): One NicoDerm CQ patch once daily for first 6 weeks (42 days). Dosage will taper from 21 mg (Weeks 1-3) to 14 mg (Weeks 4-5) to 7 mg (Week 6).
  Brief Supportive and Behavioral Treatment: Brief, standard, manualized individual cognitive behavioral therapy intervention will be based on the Freedom from Smoking curriculum from the American Lung Association.
Arm/Group | EVP-6124 + NicoDerm CQ (Active) | EVP-6124 + NRT Patch (Placebo) | Placebo + NicoDerm CQ (Active) | Placebo + NRT Patch (Placebo)
Number analyzed (Participants) | 40 | 41 | 38 | 41
% participants with 7-Day Point Prevalen
  Seven-Day Point Prevalence Abstinence Rate week 1 | 25.0 | 12.2 | 28.9 | 17.1
  Seven-Day Point Prevalence Abstinence Rate week 2 | 47.5 | 19.5 | 42.1 | 24.4
  Seven-Day Point Prevalence Abstinence Rate week 4 | 40.0 | 17.1 | 44.7 | 19.5
  Seven-Day Point Prevalence Abstinence Rate week 6 | 52.5 | 14.6 | 34.2 | 22.0
  Seven-Day Point Prevalence Abstinence Rate week 8 | 37.5 | 14.6 | 28.9 | 24.4
  Seven-Day Point Prevalence Abstinence Rate week 10 | 37.5 | 12.2 | 23.7 | 24.4
  Seven-Day Point Prevalence Abstinence Rate week 12 | 25.0 | 12.2 | 18.4 | 19.5

2. Primary Outcome: Difference in Expired Carbon Monoxide (CO) Concentration From Baseline to End Point
Description: CO concentration was measured at every visit.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 10, 12
Measure: Mean (Standard Deviation); unit: part per million
Arm/Group | EVP-6124 + NicoDerm CQ (Active) | EVP-6124 + NRT Patch (Placebo) | Placebo + NicoDerm CQ (Active) | Placebo + NRT Patch (Placebo)
Number analyzed (Participants) | 40 | 41 | 38 | 41
part per million
  Baseline | 20.2 (11) | 17.2 (9.8) | 20.5 (13.7) | 19.3 (9.4)
  Week 1 | 8.6 (11) | 9.2 (10.1) | 5.2 (6) | 8.1 (8.6)
  Week 2 | 7.7 (11.5) | 10.1 (10.2) | 4.9 (5.4) | 8.5 (8.5)
  Week 4 | 6.1 (7.7) | 9.8 (11.5) | 6.3 (7.9) | 9.6 (10.5)
  Week 6 | 7.5 (11.4) | 12.7 (16.3) | 5.3 (5.7) | 7.8 (6.4)
  Week 8 | 7.2 (10.5) | 12.6 (16.8) | 7.5 (6.4) | 7.6 (6.8)
  Week 10 | 7.2 (10.9) | 11.2 (11.9) | 8.2 (7.4) | 5.3 (5)
  Week 12 | 8.8 (8.7) | 11.4 (13.6) | 9 (8.1) | 8.3 (9.3)

3. Secondary Outcome: Effects of EVP-6124 on Cognitive Performance as Measured by the Continuous Performance Test Hit Reaction Time
Description: The Continuous Performance Test (CPT) is a measure of both vigilance/attentional control and response inhibition. During the task, subjects are required to press a button whenever a letter appears on the screen unless that letter is an 'X'. Measures of attentional control will serve as primary measure from this test. Baseline attentional impairment is associated with reduced odds of abstinence, abstinence differentially worsens performance on this measure in those with baseline attentional impairment, and NRT improves performance on a similar measure.
Time Frame: Baseline, week 1, week 12
Measure: Mean (Standard Deviation); unit: mili seconds
Arm/Group | EVP-6124 + NicoDerm CQ (Active) | EVP-6124 + NRT Patch (Placebo) | Placebo + NicoDerm CQ (Active) | Placebo + NRT Patch (Placebo)
Number analyzed (Participants) | 40 | 41 | 38 | 41
mili seconds
  Baseline Hit RT | 436.26 (78.15) | 434.72 (65.40) | 427.76 (66.87) | 423.94 (72.58)
  Week 1 Hit RT | 424.77 (76.85) | 429.99 (59.94) | 418.74 (60.32) | 407.97 (68.01)
  Week 12 Hit RT | 441.73 (71.59) | 421.66 (67.67) | 432.56 (73.91) | 396.78 (53.44)

4. Secondary Outcome: Safety and Tolerability of EVP-6124 Alone or Combined With NRT
Description: All AEs (adverse experiences) spontaneously reported by subjects and/or observed by investigator and evaluation of physical examinations, prior and concomitant medications, clinical laboratory tests, ECGs, and vital signs measurements. Data was collected at every visit and was analyzed as aggregate at the end of week 12
Time Frame: Weeks 1-12
Measure: Count of Participants; unit: Participants
Arm/Group | EVP-6124 + NicoDerm CQ (Active) | EVP-6124 + NRT Patch (Placebo) | Placebo + NicoDerm CQ (Active) | Placebo + NRT Patch (Placebo)
Number analyzed (Participants) | 40 | 41 | 38 | 41
Participants | 35 | 30 | 34 | 34

5. Secondary Outcome: Effects of EVP-6124 on Working Memory as Measured by the N-Back Task Reaction Time
Description: This task is a standard measure that can assess working memory performance under varying levels of task demand. Subjects are presented with a stream of stimuli, and the task is to decide for each stimulus whether it matches the one presented N items before. The processing load can be varied systematically by manipulating the value of N, which is expressed with changes in accuracy and reaction time. The number of errors as well as reaction times increase monotonically with increasing levels of N. The n-back task is sensitive to nicotine administration and abstinence effects. Here we present reaction time (RT)
Time Frame: Baseline, week 1, week 12
Measure: Mean (Standard Deviation); unit: mili seconds
Arm/Group | EVP-6124 + NicoDerm CQ (Active) | EVP-6124 + NRT Patch (Placebo) | Placebo + NicoDerm CQ (Active) | Placebo + NRT Patch (Placebo)
Number analyzed (Participants) | 40 | 41 | 38 | 41
mili seconds
  Baseline 2-Back RT | 634.04 (166.51) | 645.01 (180.83) | 632.80 (176.78) | 616.33 (186.83)
  Baseline 3-Back RT | 667.75 (202.35) | 642.89 (182.20) | 620.55 (210.04) | 600.78 (179.64)
  Week 1 2-Back RT | 578.58 (101.86) | 619.42 (174.86) | 565.84 (148.24) | 553.90 (135.00)
  Week 1 3-Back RT | 635.08 (164.16) | 627.85 (180.06) | 608.94 (152.38) | 586.15 (173.28)
  Week 12 2-Back RT | 608.03 (145.92) | 620.28 (175.61) | 598.47 (156.28) | 565.41 (149.08)
  Week 12 3-Back RT | 639.51 (175.91) | 613.75 (176.40) | 611.85 (185.75) | 585.15 (177.86)

ADVERSE EVENTS:
Time Frame: week 1 to week 12
Arm/Group | EVP-6124 + NicoDerm (Active) | EVP-6124 + NRT Patch (Placebo) | Placebo + NicoDerm (Active) | Placebo + NRT Patch (Placebo)
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/41 | 1/38 | 0/41
Other Adverse Events (participants affected / at risk) | 35/40 | 30/41 | 34/38 | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVP-6124 + NicoDerm (Active) (N=40) | EVP-6124 + NRT Patch (Placebo) (N=41) | Placebo + NicoDerm (Active) (N=38) | Placebo + NRT Patch (Placebo) (N=41)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis Flare (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVP-6124 + NicoDerm (Active) (N=40) | EVP-6124 + NRT Patch (Placebo) (N=41) | Placebo + NicoDerm (Active) (N=38) | Placebo + NRT Patch (Placebo) (N=41)
Constipation (Gastrointestinal disorders) | 11 (11) | 8 (8) | 8 (8) | 5 (5)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (4) | 7 (7) | 7
Elevated Creatine phosphokinase (CPK) (General disorders) | 2 (2) | 0 (0) | 4 (4) | 3 (3)
Depressive symptoms (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Headache (General disorders) | 10 (10) | 2 (2) | 2 (2) | 4 (4)
Cold/flu (Infections and infestations) | 7 (7) | 3 (3) | 7 (7) | 3 (3)
Skin Irritation at Patch Site (Skin and subcutaneous tissue disorders) | 12 (12) | 3 (3) | 2 (2) | 3 (3)
Fatigue (General disorders) | 5 (5) | 2 (2) | 2 (2) | 2 (2)
Insomnia (General disorders) | 6 (6) | 3 (3) | 6 (6) | 5 (5)
Stomach pain (Gastrointestinal disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Nausea (General disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
weight gain (General disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Irritability (General disorders) | 4 (4) | 1 (1) | 1 (1) | 3 (3)
Increase appetite (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2) | 0 (0) | 1 (1)
Allergies (General disorders) | 6 (6) | 2 (2) | 3 (3) | 3 (3)
Abnormal sleeping pattern (General disorders) | 5 (5) | 1 (1) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No